CLINICAL TRIAL: NCT05719727
Title: Prevalence and Clinicopathologic Pattern of Primary Eosinophilic Colitis in Symptomatic Patients.
Brief Title: Primary Eosinophilic Colitis in Symptomatic Patients.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa M.Abokresha, Lecturer of gastroenterology and hepatology, Assiut University
Other Study IDs: Esinophilic colitis
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Eosinophilic Colitis
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: colonoscopy — lower colonoscopy

SUMMARY:
The aim of the present study was to know the prevalence of primary eosinophilic colitis(PEC) in patients with lower gastrointestinal symptoms including diarrhea and chronic abdominal pain for which no other causes were identified.

DETAILED DESCRIPTION:
The presence of eosinophils in the different segments of the digestive tract is common and seen in diverse clinical scenarios. Eosinophilic gastrointestinal diseases (EGIDs) are a group of disorders characterized by symptoms of gastrointestinal dysfunction, caused by the inflammatory infiltration of eosinophils and include eosinophilic esophagi-tis, eosinophilic gastroenteritis, and eosinophilic colitis.

Primary eosinophilic colitis (PEC) is defined as an inflammatory disease of unknown etiology that mainly manifests as abdominal pain and diarrhea, segmental or diffuse infiltration of eosinophils in the mucosa of the colon, for which other possible causes have been ruled out .

The usual endoscopic findings tend to be nonspecific, and even though PEC is considered a rare disease, its prevalence is unknown. Evaluation of the colonic mucosa is very helpful in detecting inflammatory bowel disease, ischemic colitis, microscopic colitis ,neoplasia, and intraepithelial infections.

The endoscopic appearance of the colon is normal, or almost normal, in some of those diseases, and thus they can go by undetected

ELIGIBILITY:
Inclusion Criteria:

* All in- patients and out- patients above 18 y old undergo colonoscopy unit in Al Raghy hospital with unexplained lower symptoms including abdominal pain ,diarrhea, IBS predominant diarrhea, between , between February 2023 and December 2024 and

Exclusion Criteria:

* Cases diagnosed with 2ry causes for colonic eosinophilia.
* Patients with a known or compensated organic disease associated with diarrhea and alarm features (e.g., involuntary weight loss > 10% of the baseline weight, within the past 6 months.
* Patients with anemia, cancer and history of organ transplantation.
* Patients with HIV-AIDS infection.
* Patients under regular treatment with clozapine, carba-mazepine, rifampin, tacrolimus, gold salts, or non steroidal anti-inflammatory drugs, for 6 months prior to disease onset.
* Patients contraindicated for colonoscopy or biopsy, and patients with incomplete colonoscopy or inadequate bowel cleanliness at the time of the study .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients will be subjected to :
  1. Detailed history, clinical examination
  2. Laboratory tests :
     I-CBC, ESR or CRP or both, ,complete stool analysis . II- Fecal occult blood, fecal calprotectin when indicated in selected patients. III- Autoimmune antibody including ANA,antiDNA ,ANCA,ASCA when indicated in selected patients .
  3. CT imaging when indicated
  4. COLONOSCOPY examination :
  All patients underwent colonoscopy with random biopsies of all the colonic segments (at least 10 biop-sies per study,even in the presence of normal-appearing mucosa, and had biopsies of the segments with minimal alterations (areas oferythema, with hemorrhagic spots, loss of vascular pattern,and a nodular appearance, among others) At El-Raghy colonoscopy unit , Assuit university hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of PEC in patients with lower gastrointestinal symptoms including diarrhea and chronic abdominal pain for which no other causes were identified. | Baseline
  Estimation the prevalence of eosinophilic colitis

CONTACTS AND LOCATIONS:
Overall Officials: Hussein A elamin, MD, Study Director — Pro. Internal medicine and gastroentrology and hepatology unit; Hyam Fathy, MD, Study Chair — consultant of internal medicine gastroentrology and hepatology unit

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Egan M, Furuta GT. Eosinophilic gastrointestinal diseases beyond eosinophilic esophagitis. Ann Allergy Asthma Immunol. 2018 Aug;121(2):162-167. doi: 10.1016/j.anai.2018.06.013. Epub 2018 Jun 22. PMID 29940308
- [Result] Villanueva MS, Alimi Y. Microscopic colitis (lymphocytic and collagenous), eosinophilic colitis, and celiac disease. Clin Colon Rectal Surg. 2015 Jun;28(2):118-26. doi: 10.1055/s-0035-1549365. PMID 26034409
- [Result] Impellizzeri G, Marasco G, Eusebi LH, Salfi N, Bazzoli F, Zagari RM. Eosinophilic colitis: A clinical review. Dig Liver Dis. 2019 Jun;51(6):769-773. doi: 10.1016/j.dld.2019.04.011. Epub 2019 May 20. PMID 31122823